CLINICAL TRIAL: NCT01985581
Title: A Single-Center, Randomized, Double Blind, Placebo-Controlled, Crossover Evaluation of the Effect of GXR as Adjunctive Treatment With Stimulant on Executive Function and Quality of Life at Home and School in Children With ADHD
Brief Title: Efficacy of GXR as Adjunctive Therapy With Psycho-stimulant on Executive Function in Children With ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JPM van Stralen Medicine Professional (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RES 13-001
Record Dates: First submitted 2013-10-27; First posted 2013-11-15 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; Intuniv extended release; Executive Function; Quality of Life
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo first then GXR (Experimental): patient will continue to take stable dosage of usual stimulant therapy (Ritalin, Ritalin SR, Biphentin, Concerta, Vyvanse, Adderall or Dexedrine). In the first intervention period subject took placebo and second intervention period subject took GXR. GXR dose was optimized to between 1 and 4mg.
  Interventions: Drug: Guanfacine extended release; Drug: Placebo; Drug: Stimulant therapy
- GXR first then Placebo (Placebo Comparator): patient will continue to take stable dosage of usual stimulant(Ritalin, Ritalin SR, Biphentin, Concerta, Vyvanse, Adderall or Dexedrine). In the first intervention period subject took GXR and second intervention period subject took placebo. GXR dose was optimized to between 1 and 4mg.
  Interventions: Drug: Guanfacine extended release; Drug: Placebo; Drug: Stimulant therapy

INTERVENTIONS:
Drug: Guanfacine extended release
  Other Names: Intuniv extended release
Drug: Placebo
Drug: Stimulant therapy — patient will continue to take stable dosage of usual stimulant therapy (Ritalin, Ritalin SR, Biphentin, Concerta, Vyvanse, Adderall or Dexedrine)

SUMMARY:
This study looks to examine whether or not INTUNIV extended release can help children aged 6-12 years diagnosed with Attention-Deficit/Hyperactivity Disorder (ADHD) in improving Executive Function when added to their usual care stimulant therapy. Executive functions are a set of mental processes that include emotional control, planning, organization, working memory, inhibition of behaviors, and managing time and space. As children with ADHD usually have difficulties with Executive Function, and Executive function difficulties lead to more difficulties in school and behaviour, it is anticipated that adding INTUNIV extended release to usual stimulant therapy will improve Executive Function scores as rated by parents and teachers. Improvements in quality of life will also be measured.

DETAILED DESCRIPTION:
Although stimulant medications have been shown to have positive impact on executive function (EF) (Findling et al, 2009; Hale et al. 2011), little has been documented about the effect of INTUNIV extended release on EF in children. The manifestation of clinical symptoms related to impairment in EF often leads to the search for additional treatment options and in many cases to adjunct therapies to the traditional stimulant medication treatment regimen. Demonstrating that the addition of INTUNIV extended release to usual stimulant therapy is effective for symptom control as well as in improving EF may influence clinical treatment algorithms and the need for health care resources to effectively manage patients. Since EF deficits negatively impact academic achievement and behavior at school and because children spend a large number of daytime hours at school, the concordance of any reported improvement in the school and the home environment will be examined. Overall improvement in quality of life with the addition of INTUNIV extended release will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient aged 6 to 12 years at the time of consent/assent and to then of study. A patient who would turn 13 before the end of the study cannot be enrolled
2. Patient's parent or legally authorized representative (LAR) must provide signed informed consent before any study-related procedures are completed.
3. Patient meets the diagnostic standard manual-5 criteria for a primary diagnosis of ADHD, combined sub-type, hyperactive/impulsive sub-type, or inattentive sub-type
4. Patient is currently on a stable stimulant regimen but whose EF is suboptimal. Suboptimal EF is defined as a global executive composite t-score greater than 65 (>1.5 SD from mean) on the BRIEF-P questionnaire at screening.
5. Patient who is currently and is expected to remain on a stable stimulant regimen throughout the study. A stable stimulant regimen is defined as:

   •No significant change in dose or dosing frequency within the past 30 days prior to screening and stimulant is felt to be optimized by the investigator.
6. Patient is functioning at an age-appropriate level intellectually, as judged by the Investigator.
7. Patient is able to swallow intact tablets.
8. Patient has sitting blood pressure (BP) measurement within the 95th percentile for age, sex, and height (see Blood Pressure Levels for Boys and Girls by Age and Height Percentile
9. Patient and parent/LAR understand, are willing, able, and likely to fully comply with the study procedures and restrictions defined in this protocol.

Exclusion Criteria:

1. Patient has a current, controlled (requiring a prohibited medication or behavioural modification program) or uncontrolled, co-morbid psychiatric diagnosis [except oppositional defiant disorder (ODD)], including any severe co-morbid Axis II disorders or severe Axis I disorders such as post-traumatic stress disorder (PTSD), bipolar illness, psychosis, pervasive developmental disorder, obsessive-compulsive disorder (OCD), substance abuse disorder, or other symptomatic manifestations or lifetime history of bipolar illness, psychosis or conduct disorder.
2. Patient has any condition or illness which, in the opinion of the Investigator, represents an inappropriate risk to the patient and/or could confound the interpretation of the study. Mild stable asthma treated without the use of beta-2 agonist is not exclusionary.
3. Patient has a known personal history, or presence, of structural cardiac abnormalities, cardiovascular or cerebrovascular disease, serious heart rhythm abnormalities, syncope, tachycardia, cardiac conduction problems (e.g., clinically significant heart block or QT interval prolongation: QTc >0.44 seconds), exercise-related cardiac events including syncope and pre-syncope, or clinically significant bradycardia.
4. Patient has a known family history (in siblings, parents, and/or grand-parents) of sudden cardiac death, ventricular arrhythmia, or QT prolongation (QTc >0.44 seconds).
5. Patient has a known history of hypertension (see Blood Pressure Levels for Boys and Girls by Age and Height Percentile
6. Patient has glaucoma.
7. Patient has a history of a seizure disorder (other than a simple childhood febrile seizure).
8. Patient has renal or hepatic insufficiency
9. Patient is currently using prohibited medication.
10. Patient has taken another investigational product within 30 days prior to the Enrolment Visit.
11. Patient has a known or suspected allergy, hypersensitivity, or clinically significant intolerance to guanfacine hydrochloride or any of its active ingredients or patient is taking other products containing guanfacine.
12. History of adverse event or failure to respond (lack of efficacy) to an adequate trial of an alpha-agonist.
13. Patient is female and is pregnant or currently lactating.
14. Patient is currently considered a suicide risk in the opinion of the Investigator, has previously made a suicide attempt, or has a prior history of, or is currently demonstrating active suicide ideation. Patients with intermittent passive suicidal ideation are not necessarily excluded based on the assessment of the Investigator.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2013-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judy PM van Stralen, MD, Principal Investigator — JPM van Stralen Medicine Professinal Organization
Locations (1):
- JPM van Stralen Medicine Professional Corporation, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from principal investigators clinical practice as well as through advertisement in local medical offices and through print and radio advertisements
Groups:
- Placebo First Then GXR: patient will continue to take stable dosage of usual stimulant therapy (Ritalin, Ritalin SR, Biphentin, Concerta, Vyvanse, Adderall or Dexedrine) and placebo for the first intervention period and GXR for the second intervention period (after a washout period). GXR dose was optimized to between 1 and 4mg.
- GXR First Then Placebo: patient will continue to take stable dosage of usual stimulant therapy (Ritalin, Ritalin SR, Biphentin, Concerta, Vyvanse, Adderall or Dexedrine) and GXR for the first intervention period and placebo for the second intervention period (after a washout period). GXR dose was optimized to between 1 and 4mg.
Period: First Intervention
Arm/Group | Placebo First Then GXR | GXR First Then Placebo
Started | 25 | 25
Completed | 22 | 23
Not Completed | 3 | 2
Period: Second Intervention
Arm/Group | Placebo First Then GXR | GXR First Then Placebo
Started | 22 | 23
Completed | 20 | 19
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- PLB First Then GXR: subjects received PLB in first arm of study and GXR in second arm. subject continued to take stable dosage of usual stimulant therapy (Ritalin, Ritalin SR, Biphentin, Concerta, Vyvanse, Adderall or Dexedrine)
- GXR First Then PLB: subjects received GXR in first arm of study and PLB in second arm subject continued to take stable dosage of usual stimulant therapy (Ritalin, Ritalin SR, Biphentin, Concerta, Vyvanse, Adderall or Dexedrine)
- Total: Total of all reporting groups
Arm/Group | PLB First Then GXR | GXR First Then PLB | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Median (Full Range); unit: years] | 9.0 [7 to 11] | 10 [7 to 12] | 9.5 [7 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 20 | 22 | 42
Region of Enrollment [Number; unit: participants]
  Canada | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Effect of Adjunctive INTUNIV Extended Release Treatment on Executive Function as Assessed by Change From Baseline on the BRIEF-parent Questionnaires
Description: The Behavioural Rating Inventory of Executive Function (BRIEF) was developed to assess such real-world expressions of executive function in the home (BRIEF-P) as assessed by the parent. This is an 86 item questionnaire completed by the parents. The score is converted to a t-score with a score less than 65 being considered within the normal range. Higher scores are worsening in function.
Time Frame: measured at baseline and end of each 12 week treament arm
Population: ITT population - consisting of subjects who took at least one dose of treatment and completed at least one non-baseline BRIEF questionnaire during either period 1 or period 2.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo and Stimulant: Subjects received placebo and usual stimulant therapy
- GXR and Stimulant: Subjects received GXR (1-4 mg as optimized dosage) in addition to usual stimulant therapy
Arm/Group | Placebo and Stimulant | GXR and Stimulant
Number analyzed (Participants) | 48 | 47
units on a scale | -5.3 (1.46) | -6.9 (1.53)
Statistical Analysis 1: Comparison: Placebo and Stimulant vs GXR and Stimulant; Test type: Superiority or Other; p = 0.0392, ANOVA; LS mean difference = -3.0, 95% CI 2-sided [-5.9 to -0.2]

2. Secondary Outcome: Effect of Adjunctive INTUNIV Extended Release Treatment on Change in Quality of Life as Assessed by the KINDL®-Child Questionnaire.
Description: The KINDL is a quality of life questionnaire of 24 items completed by the subject (KINDL-child). It is a generic instrument for assessing Health Related quality of life in children and adolescents aged 3 years and older. Norm values are given based on representative German data from the German National Health Interview and Examination Survey for Children and Adolescents (KiGGS) study, a broad survey realized by the German Robert-Koch Institute. The KINDL scores were converted to range between 0 and 100 with higher scores indicating better quality of life as reported by the child
Time Frame: Measured at baseline and end of each 12 week treatment arm
Population: ITT population - consisting of subjects who took at least one dose of treatment and completed at least one non-baseline questionnaire during either period 1 or period 2.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo and Stimulant: The quality of life was measured in those patients taking placebo along with their usual stimulant therapy
- GXR and Stimulant: The quality of life was measured in those patients taking GXR along with their usual stimulant therapy
Arm/Group | Placebo and Stimulant | GXR and Stimulant
Number analyzed (Participants) | 47 | 46
units on a scale | 0.8 (1.58) | 1.2 (1.62)
Statistical Analysis 1: Comparison: Placebo and Stimulant vs GXR and Stimulant; Test type: Superiority or Other; p = 0.894, ANOVA; LS mean difference = 0.3, 95% CI 2-sided [-4.0 to 4.6]

3. Secondary Outcome: Effect of Adjunct Therapy on ADHD Symptom Control as Assessed by the Change in the ADHD Rating Scale (ADHD-RS-IV)
Description: The ADHD-RS-IV is completed by the Investigator familiar with the scale. It is an 18 item scale designed to reflect current symptomatology of ADHD based on the DSM-5 criteria. Each item is scored from a range of 0 (reflecting no symptoms) to 3 (reflecting severe symptoms) with total scores ranging from 0-54, with higher scores reflecting more severe symptoms
Time Frame: comparison from baseline to end of each 12 week treatment arm
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo and Stimulant: subjects continued to take usual dose stimulant and took placebo
- GXR and Stimulant: Patients continued to take usual dose stimulant and optimized dose (1-4mg) of GXR
Arm/Group | Placebo and Stimulant | GXR and Stimulant
Number analyzed (Participants) | 48 | 47
units on a scale | -5.5 (1.63) | -11.1 (1.51)
Statistical Analysis 1: Comparison: Placebo and Stimulant vs GXR and Stimulant; Test type: Superiority or Other; p = 0.0001, ANOVA; LS mean difference = -6.2, 95% CI 2-sided [-9.1 to -3.2]

4. Secondary Outcome: Subjects Experiencing Suicidal Ideation, Suicidal Behaviour and Self-injurious Behaviour Without Suicidal Intent and Incident of Serious Adverse Events in Each Treatment Arm
Description: To compare the number of subjects experiencing suicidal ideation, suicidal behaviour and self-injurious behaviour without suicidal intent as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) and incident of Serious Adverse Events (SAEs) in each treatment arm
Time Frame: Measured up to 30 weeks
Population: as for outcome 2
Measure: Number; unit: subjects
Groups:
- Stimulant & Placebo: patient will continue to take stable dosage of usual stimulant(Ritalin, Ritalin SR, Biphentin, Concerta, Vyvanse, Adderall or Dexedrine)therapy plus placebo
  Placebo
- Stimulant and Guanfancine Extended Release: patient will continue to take stable dosage of usual stimulant therapy (Ritalin, Ritalin SR, Biphentin, Concerta, Vyvanse, Adderall or Dexedrine) and also receive guanfacine extended release at a individually optimized dosage of 1-4 mg.
  Guanfacine extended release
Arm/Group | Stimulant & Placebo | Stimulant and Guanfancine Extended Release
Number analyzed (Participants) | 50 | 50
subjects | 1 | 1

5. Secondary Outcome: Evaluate the Effect of Adjunctive INTUNIV Extended Release Treatment on Change in Quality of Life as Assessed by the KINDL®-Parent Questionnaire.
Description: The KINDL is a quality of life questionnaire of 24 items completed by the parent (KINDL-parent). It is a generic instrument for assessing Health Related quality of life in children and adolescents aged 3 years and older. Norm values are given based on representative German data from the German National Health Interview and Examination Survey for Children and Adolescents (KiGGS) study, a broad survey realized by the German Robert-Koch Institute. The KINDL scores were converted to range between 0 and 100 with higher scores indicating better quality of life as reported by the parent.
Time Frame: Measured at baseline and end of each 12 week treatment arm
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo and Stimulant: The child's quality of life as assessed by the parent was measured in subjects taking usual stimulant and placebo
- GXR and Stimulant: The child's quality of life as assessed by the parent was measured in subjects taking usual stimulant and GXR (optimized dose 1-4 mg)
Arm/Group | Placebo and Stimulant | GXR and Stimulant
Number analyzed (Participants) | 48 | 47
units on a scale | 3.4 (1.46) | 1.4 (1.45)
Statistical Analysis 1: Comparison: Placebo and Stimulant vs GXR and Stimulant; Test type: Superiority or Other; p = 0.8706, ANOVA; LS mean difference = 0.3, 95% CI 2-sided [-3.2 to 3.7]

6. Secondary Outcome: Effect of Adjunct Therapy on ADHD Symptom Control as Assessed by the Change on the Clinical Global Impression of Severity (CGI-S) Scale
Description: The Clinical Global Impression- Severity scale is a scale of illness ranging from 1 (normal) to 7 (among the most severely ill patients). Subjects who felt normal, not at all ill or borderline mentally ill are considered improved. The outcome measure is reporting the percentage of participants showing improvement
Time Frame: comparison from baseline to end of each 12 week treatment arm
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Groups:
- Placebo and Stimulant: subjects who continued to take usual stimulant dosage and took placebo
- GXR and Stimulant: subjects who continued to take usual stimulant dosage and took GXR at optimized dose of 1-4 mg
Arm/Group | Placebo and Stimulant | GXR and Stimulant
Number analyzed (Participants) | 48 | 47
percentage of subjects | 10.6 | 29.8

7. Secondary Outcome: Evaluate the Effect of Adjunct Therapy on ADHD Symptom Control as Assessed by the Change in Clinical Global Impression of Improvement (CGI-I) Scale
Description: CGI-I is a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Subjects who felt very much improved or much improved are considered improved.The outcome measure is reporting the percentage of participants showing improvement
Time Frame: comparison from baseline to end of each 12 week treatment arm
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Groups:
- GXR and Stimulant: subjects who continued to take usual stimulant dosage and took GXR (optimized dose 1-4 mg)
Arm/Group | Placebo and Stimulant | GXR and Stimulant
Number analyzed (Participants) | 48 | 47
percentage of subjects | 27.7 | 57.4

ADVERSE EVENTS:
Time Frame: from time consent was signed until end of study (week 30)
Groups:
- Stimulant and GXR: adverse event frequency in those taking stimulant + GXR
- Stimulant and PLB: adverse event frequency in those taking stimulant + PLB
Arm/Group | Stimulant and GXR | Stimulant and PLB
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/48
Other Adverse Events (participants affected / at risk) | 41/47 | 41/48
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stimulant and GXR (N=47) | Stimulant and PLB (N=48)
Headache (Nervous system disorders) | 23 | 16
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 12 | 18
Abdominal Upper Pain (Gastrointestinal disorders) | 14 | 5
Insomnia (Nervous system disorders) | 5 | 9
Vomiting (Gastrointestinal disorders) | 5 | 8
Fatigue (Nervous system disorders) | 11 | 1
Gastroenteritis (Gastrointestinal disorders) | 6 | 5
Affect Lability (Psychiatric disorders) | 6 | 1
Somnolence (Nervous system disorders) | 5 | 2
Pyrexia (General disorders) | 3 | 3
Nauseau (Gastrointestinal disorders) | 1 | 4
Sleep disorder (General disorders) | 3 | 1

LIMITATIONS AND CAVEATS:
There was insufficient teacher data collected to interpret the results. Children appeared to struggle with the completion of the KINDL calling in to question the validity of the results of this questionnaire

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No